CLINICAL TRIAL: NCT05253053
Title: A Phase Ib/II Study of TT-00420 Tablet, as Monotherapy or in Combination Regimens, to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy in Patients With Advanced Solid Tumor
Brief Title: To Evaluate Efficacy and Safety of TT-00420 (Tinengotinib) as Monotherapy and Combination Therapy in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TransThera Sciences (Nanjing), Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TT00420CN04
Record Dates: First submitted 2022-01-26; First posted 2022-02-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumor; Cholangiocarcinoma; Biliary Tract Cancer; HER2-negative Breast Cancer; Triple Negative Breast Cancer; Small-cell Lung Cancer; Bladder Cancer; Prostate Cancer; Thyroid Cancer; Gastric Cancer; Gallbladder Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms; Triple Negative Breast Neoplasms; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms; Prostatic Neoplasms; Thyroid Neoplasms; Stomach Neoplasms; Gallbladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Study will consist of three arms: Arm A (TT-00420 Tablet Monotherapy), Arm B (TT-00420 tablet in combination with atezolizumab(Tecentriq®)) and Arm C (TT-00420 tablet in combination with nab-paclitaxel (Abraxane®)).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: TT-00420 Tablet Monotherapy (Experimental): TT-00420 tablets will be administered once daily in 21-day cycles. Dose escalation will be guided by a 3+3 design in Phase Ib to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: TT-00420
- Arm B: TT-00420 tablet in combination with Atezolizumab Injection (Tecentriq ®) (Experimental): TT-00420 tablets will be administered once daily in 21-day cycles. Atezolizumab(1200 mg/20 mL) will be administered intravenously on Day 1 of each 21-day cycle. Dose escalation will be guided by a 3+3 design in Phase Ib to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: TT-00420; Drug: Combination Product: Atezolizumab
- Arm C: TT-00420 tablet in combination with nab-paclitaxel (Abraxane®) (Experimental): TT-00420 tablets will be administered once daily in 21-day cycles. Nab-paclitaxel 125 mg/m^2 will be administered intravenously on Day 1 and 8 of each 21-day cycle. Dose escalation will be guided by a 3+3 design in Phase Ib to determine the recommended phase 2 dose (RP2D).
  Interventions: Drug: TT-00420; Drug: Combination Product: Nab-Paclitaxel

INTERVENTIONS:
Drug: TT-00420 — TT-00420 tablet will be administered orally once daily per protocol defined schedule.
Drug: Combination Product: Atezolizumab — Atezolizumab would be administered via infusion on Day 1 of 21-day cycle
  Arms: Arm B: TT-00420 tablet in combination with Atezolizumab Injection (Tecentriq ®)
Drug: Combination Product: Nab-Paclitaxel — Nab-Paclitaxel would be administered via infusion on Day 1 and 8 of 21-day cycle
  Arms: Arm C: TT-00420 tablet in combination with nab-paclitaxel (Abraxane®)

SUMMARY:
This is a Phase Ib/II, multicenter, open-label study to evaluate the safety and preliminary efficacy of TT-00420 tablet, as monotherapy or in combination regimens, in patients with advanced solid tumors (solid tumor, BTC and TNBC).

DETAILED DESCRIPTION:
Study consists of three arms, Arm A is a Phase Ib/II study of TT-00420 tablet monotherapy, Arm B is a Phase Ib/II study of TT-00420 tablet in combination with atezolizumab (Tecentriq®), and Arm C is a Phase Ib/II study of TT-00420 tablet in combination with nab-paclitaxel (Abraxane®).

Arm A: TT-00420 Tablet Monotherapy Phase Ib will enroll patients with preferred indications including advanced cholangiocarcinoma, small cell lung cancer, HER2-negative breast cancer including TNBC, bladder cancer, prostate cancer, thyroid cancer, gastric cancer, gallbladder cancer and other advanced solid tumors to receive TT-00420 monotherapy. Phase Ib will be a dose escalation study of TT-00420 in combination, guided by 3+3 design, to determine a Recommended Phase 2 Dose (RP2D). Based on preliminary efficacy results, Phase II will enroll additional patients in select indications to evaluate the efficacy of TT-00420 monotherapy.

Arm B: TT-00420 tablet in combination with atezolizumab (Tecentriq®) Arm B will enroll patients with advanced biliary tract cancer. Phase Ib will be a dose escalation study of TT-00420 in combination with nab-paclitaxel, guided by 3+3 design, to determine a Recommended Phase 2 Dose (RP2D). Phase II will enroll additional patients with advanced biliary tract cancer to further evaluate the efficacy of the combination regimen.

Arm C: TT-00420 tablet in combination with nab-paclitaxel (Abraxane®) Arm C will enroll patients with advanced triple-negative breast cancer (TNBC). Phase Ib will be a dose escalation study of TT-00420 in combination with nab-paclitaxel, guided by 3+3 design, to determine a Recommended Phase 2 Dose (RP2D). Phase II will enroll additional patients with advanced TNBC to further evaluate the efficacy of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Arm A：Histopathological or cytologically documented locally advanced or metastatic and solid tumors（including but not limited to advanced cholangiocarcinoma, small cell lung cancer, HER2-negative breast cancer including TNBC, bladder cancer, prostate cancer, thyroid cancer, gastric cancer, gallbladder cancer and other advanced solid tumors.

   Arm B：Histopathological or cytologically documented locally advanced or metastatic and Unresectable advanced biliary tract malignant tumors (except ampullary carcinoma).

   Arm C：
   * Histopathological invasive advanced TNBC with triple-negative receptor status that meets the institution standards was proved ER or PR by IHC (positive tumor nucleus<10% )
   * HER2-negative (ASCO-CAP guideline [Wolff A C, 2018] )
3. Received all currently available standard treatments (unless the treatment is contraindicated, intolerable, or unavailable for any reason)
4. At least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. 6. Adequate organ and bone marrow function(without receiving any hematopoietic growth factor, blood or platelet therapy within 1 week before the first dose.

   * Complete blood count (CBC):

     * Absolute Neutrophil Count (ANC)≥ 1.5 × 109/L
     * Hemoglobin（Hgb）≥ 9 g/dl
     * Platelets（Plt）≥ 75 × 109/L
   * Liver function:

     * AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 × ULN if liver metastases are present .
     * Total bilirubin ≤ 1.5 × ULN or direct bilirubin<ULN (if total bilirubin>1.5 ULN).
     * Patients with hepatocellular carcinoma (HCC) and BTC: Child Pugh A or B (Score ≤ 7).
   * Renal fuction:

     * serum creatinine ≤ 1.5 × ULN or Calculated 24-hour clearance ≥ 50 mL/min (Cockcroft Gault formula).
7. Must agree to take sufficient contraceptive methods to avoid pregnancy during the study and until at least 6 months after ceasing study treatment
8. Able to sign informed consent and comply with the protocol

Exclusion Criteria:

Patients who meet one or more of the following criteria will not be included in this study:

1. Women who are pregnant or lactating
2. Women of child-bearing potential (WOCBP) who do not use adequate birth control
3. Patients with any hematologic malignancy, including leukemia (any form), lymphoma, and multiple myeloma
4. Patients with a history of

   * primary central nervous system tumors or
   * carcinomatous meningitis (also known as leptomeningeal disease). Note: Patients with treated brain metastases that are off corticosteroids and have been clinically stable for 28 days are eligible for enrollment.
5. Impaired cardiac function or significant diseases, including but not limited to any of the following:

   * left ventricular ejection fraction (LVEF) < 45% as determined by multigated acquisition (MUGA) scan or echocardiogram (ECHO)
   * Congenital long QT syndrome
   * QTcF ≥ 450 msec on screening ECG
   * Unstable angina pectoris ≤ 3 months prior to starting study drug
   * Acute myocardial infarction ≤ 3 months prior to starting study drug
6. Patients who are currently receiving treatment with medication that has known risk to prolong the QT interval or induce Torsades de Pointes, and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug.
7. Patients with impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of TT-00420
8. Patients who have received chemotherapy, targeted therapy, or immunotherapy ≤ 4 weeks (6 weeks for nitrosourea or mitomycin-C) prior to starting study drug or who have not recovered from side effects of such therapy
9. Patients who have undergone major surgery or wide field radiotherapy ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
10. Patients who are currently receiving treatment with strong CYP3A inhibitors or inducers ≤ 2 weeks prior to starting study drug.
11. Patients who have used of proton pump inhibitors (PPIs) within 4 days or histamine H2 blockers within 2 days prior to starting study drug
12. Human Immunodeficiency Virus (HIV) positive
13. Patients with active HBV infection (HBV DNA copy number ≥ ULN) and/or HCV infection (HCV RNA copy number ≥ ULN)
14. Patients with active tuberculosis
15. Has received a live-virus vaccination within 30 days of planned first dose Note：Seasonal flu and COVID-19 vaccines are permitted before enrollment at least 7 days.
16. Patients with a history of medical conditions, treatment, or abnormal laboratory tests that could affect the results of the study, interfere with study participation and compliance per investigator's judgment
17. 【Note】：The following three types of patients may be enrolled after being determined by the sponsor:

    ①Patients who have received emergency, low-dose, systemic immunosuppressive therapy (for example, one-time dexamethasone administration for vomiting);

    ② Patients who need steroid prophylaxis and have a history of intravenous contrast agent allergic reactions should use MRI for baseline and follow-up tumor assessment;

    ③The use of inhaled corticosteroids to treat chronic obstructive pulmonary disease, the use of mineralocorticoids (such as fludrocortisone) to treat patients with orthostatic hypotension and the use of low-dose supplementary corticosteroids to treat adrenal insufficiency are permitted.

    Arm B: TT-00420 tablet in combination with Atezolizumab Injection (Tecentriq ®): Subjects who meet one or more of the following criteria are also not allowed to participate in this study.
18. A history of severe allergies, immune stress, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
19. Known to have hypersensitivity or allergies to any ingredient of Chinese hamster ovary cells or atelizumab injection.
20. History of autoimmune diseases, including but not limited to myasthenia gravis, autoimmune myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, and antiphospholipid syndrome related Vascular thrombosis, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis or glomerulonephritis.

    【Note】The following two types of patients may be enrolled after being determined by the sponsor: ① Patients who have a history of autoimmune hypothyroidism but have stable doses of thyroid replacement hormone therapy; ② Patients who use stable doses of insulin therapy to control type I diabetes may can be enrolled.
21. Patients who have a history of allogeneic stem cell or solid organ transplantation.
22. Patients who have a history of non-specific pulmonary fibrosis, tissue pneumonia (such as: bronchiolitis obliterans, unknown tissue pneumonia), drug-induced pneumonia, or active pneumonia showed by chest CT scan.

    【Note】radiation pneumonitis (fibrosis) exist in the radiation area can be enrolled.
23. Patients who have received systemic immunostimulatory drugs therapy (including but not limited to interferon or IL-2) ≤ the shorter one of 4 weeks or 5 half-lives of immunostimulatory drugs.
24. Patients who have received systemic corticosteroids or other systemic immunosuppressive drugs (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, and Tumor Necrosis Factor (TNF)) within 2 weeks prior to starting study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | Up to 30 days from the last dose
  As assessed per NCI Common Toxicity Criteria for Adverse Events, version 5.0
Dose limiting toxicity (DLT) | Up to 21 days from the first dose
  Dose escalation cohorts are monitored and assessed using the NCI Common Toxicity Criteria for Adverse Events, version 5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an average of 9 months
  The proportion of subjects who achieved a complete response (CR) or a partial response (PR) based on RECIST version 1.1.
Disease Control Rate (DCR) | Through study completion, an average of 9 months
  Defined as CR + PR + stable disease (SD) based on RECIST version 1.1.
Duration of Objective Response (DOR) | Through study completion, an average of 9 months
  Duration of response for CR or PR based on RECIST version 1.1.
Progression Free Survival (PFS) | From first study drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall Survival (OS) | From first study drug administration until the date of death from any cause, assessed up to 24 months
Area under the curve (AUC0-∞) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 21 days)
  Blood samples will be collected at designated time points for pharmacokinetic analysis of TT-00420
Area under the curve (AUC0-t) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 21 days)
  Blood samples will be collected at designated time points for pharmacokinetic analysis of TT-00420
Maximum observed concentration (Cmax) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 21 days)
  Blood samples will be collected at designated time points for pharmacokinetic
Half-life (T1/2) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 21 days)
Time to Maximum Concentration (Tmax) | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 21 days)
Volume of Distribution | From Cycle 1 Day 1 to Cycle 2 Day 1 (each cycle is 21 days)

OTHER OUTCOMES:
Potential relationship between efficacy and biomarkers | Through study completion, an average of 9 months
  Evaluation of biomarkers, including but not limited to, FGFR2 alterations, PD-L1 expression, dMMR, MSI, TNBC subtype and TMB
changes of main circulating metabolites of TT-00420 in plasma | Through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Fudan Univisity Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No